CLINICAL TRIAL: NCT01015612
Title: CoreValve® System Australia/New Zealand Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiovascular (Industry)
Collaborators: Medtronic Australasia (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-PAVR-R2007
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic Valve Stenosis; Aortic Valve Insufficiency
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medtronic CoreValve® System Implantation (Experimental): Patients with symptomatic severe aortic stenosis who have an elevated surgical risk
  Interventions: Device: Medtronic CoreValve® System

INTERVENTIONS:
Device: Medtronic CoreValve® System — The Medtronic CoreValve® System device is designed to replace the native aortic valve without the requirement for open heart surgery and without concomitant surgical removal of the failed native valve in patients with symptomatic severe aortic stenosis who have an elevated surgical risk

SUMMARY:
To evaluate the performance, efficacy and safety of the percutaneous implantation of the CoreValve® prosthetic aortic valve in patients with severe symptomatic native aortic valve stenosis that have an elevated surgical risk

DETAILED DESCRIPTION:
Prospective, non-randomized, single-arm multi-center trial conducted under a common protocol at 10 centers in Australia and New Zealand.

ELIGIBILITY:
Inclusion Criteria

1. Documented severe aortic valve stenosis
2. Access vessel diameter >6 mm as defined pre procedure via angiographic measure
3. Aortic valve annulus diameter ≥ 20 mm and < 29 mm as defined pre procedure by echocardiographic measure
4. Ascending aorta diameter ≤ 43 mm at the sino-tubular junction
5. Native aortic valve disease, defined as valve stenosis with an aortic valve area<1cm2 (<0.6cm2 /m2) as defined pre procedure by echocardiographic measure

   AND (Assessment of Surgical Risk)

   Age ≥ 80 years

   AND/OR

   Surgical risk calculated with logistic EuroSCORE ≥ 20%,

   AND/OR

   Age ≥ 65 years with one or two (but not more than 2) of the following criteria:
   * Cirrhosis of the liver (Child class A or B)
   * Pulmonary insufficiency : VMS < 1 liter
   * Previous cardiac surgery (CABG, valvular surgery)
   * Porcelain aorta
   * Pulmonary hypertension > 60 mmHg and high probability of cardiac surgery for other than valve replacement
   * Recurrent pulmonary embolus
   * Right ventricular insufficiency
   * Thoracic burning sequelae contraindicating open chest surgery
   * History of mediastinum radiotherapy
   * Severe connective tissue disease resulting in a contraindication to surgery
   * Cachexia (clinical impression)
6. Study subjects must be willing and able to attend all follow-up visits within specified visit windows, and agree to undergo all protocol evaluations at each visit

Exclusion Criteria:

1. Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, clopidogrel, nitinol, porcine products, or contrast media which cannot be adequately pre-medicated
2. Any sepsis, including active endocarditis.
3. Recent myocardial infarction (<30 days)
4. Any left ventricular or atrial thrombus as determined pre procedure by echocardiography
5. Uncontrolled atrial fibrillation
6. Mitral or tricuspid valvular insufficiency (> grade II)
7. Previous aortic valve replacement (mechanical valve or stented bioprosthetic valve)
8. Evolutive or recent CVA (cerebrovascular accident), (<3 months)
9. Femoral, iliac or aortic vascular condition (e.g. stenosis, tortuosity), that make impossible insertion and endovascular access to the aortic valve
10. Symptomatic carotid or vertebral arteries narrowing (> 70%) disease
11. Abdominal or thoracic aortic aneurysm
12. Bleeding diathesis or coagulopathy, or patient will refuse blood transfusion
13. Evolutive disease with life expectancy less than one year
14. Creatinine clearance < 20 ml/min
15. Active gastritis or known peptic ulcer disease
16. Pregnancy

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 634 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian T Meredith, MD, Principal Investigator — Monash Heart Medical Center; Eric Vang, Study Director — Medtronic
Locations (10):
- Australia (8):
  - St. Vincents Sydney, Darlinghurst, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Hospital, Clayton, Victoria
  - St. Vincent's Melbourne, Fitzroy, Victoria
  - Epworth Hospital, Melbourne, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (2):
  - Mercy Hospital, Auckland
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonow RO, Carabello BA, Chatterjee K, de Leon AC Jr, Faxon DP, Freed MD, Gaasch WH, Lytle BW, Nishimura RA, O'Gara PT, O'Rourke RA, Otto CM, Shah PM, Shanewise JS; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2008 focused update incorporated into the ACC/AHA 2006 guidelines for the management of patients with valvular heart disease: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to revise the 1998 guidelines for the management of patients with valvular heart disease). Endorsed by the Society of Cardiovascular Anesthesiologists, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2008 Sep 23;52(13):e1-142. doi: 10.1016/j.jacc.2008.05.007. No abstract available. PMID 18848134
- [Background] Varadarajan P, Kapoor N, Bansal RC, Pai RG. Clinical profile and natural history of 453 nonsurgically managed patients with severe aortic stenosis. Ann Thorac Surg. 2006 Dec;82(6):2111-5. doi: 10.1016/j.athoracsur.2006.07.048. PMID 17126120
- [Background] Sundt TM, Bailey MS, Moon MR, Mendeloff EN, Huddleston CB, Pasque MK, Barner HB, Gay WA Jr. Quality of life after aortic valve replacement at the age of >80 years. Circulation. 2000 Nov 7;102(19 Suppl 3):III70-4. doi: 10.1161/01.cir.102.suppl_3.iii-70. PMID 11082365
- [Background] Kastrup J, Wennevold A, Thuesen L, Nielsen TT, Kassis E, Fritz-Hansen P, Thayssen P. Short- and long-term survival after aortic balloon valvuloplasty for calcified aortic stenosis in 137 elderly patients. Dan Med Bull. 1994 Jun;41(3):362-5. PMID 7924464
- [Background] Cribier A, Eltchaninoff H, Tron C, Bauer F, Agatiello C, Sebagh L, Bash A, Nusimovici D, Litzler PY, Bessou JP, Leon MB. Early experience with percutaneous transcatheter implantation of heart valve prosthesis for the treatment of end-stage inoperable patients with calcific aortic stenosis. J Am Coll Cardiol. 2004 Feb 18;43(4):698-703. doi: 10.1016/j.jacc.2003.11.026. PMID 14975485
- [Background] Cribier A, Eltchaninoff H, Tron C, Bauer F, Agatiello C, Nercolini D, Tapiero S, Litzler PY, Bessou JP, Babaliaros V. Treatment of calcific aortic stenosis with the percutaneous heart valve: mid-term follow-up from the initial feasibility studies: the French experience. J Am Coll Cardiol. 2006 Mar 21;47(6):1214-23. doi: 10.1016/j.jacc.2006.01.049. Epub 2006 Feb 9. PMID 16545654
- [Background] Grube E, Laborde JC, Gerckens U, Felderhoff T, Sauren B, Buellesfeld L, Mueller R, Menichelli M, Schmidt T, Zickmann B, Iversen S, Stone GW. Percutaneous implantation of the CoreValve self-expanding valve prosthesis in high-risk patients with aortic valve disease: the Siegburg first-in-man study. Circulation. 2006 Oct 10;114(15):1616-24. doi: 10.1161/CIRCULATIONAHA.106.639450. Epub 2006 Oct 2. PMID 17015786
- [Background] Grube E, Schuler G, Buellesfeld L, Gerckens U, Linke A, Wenaweser P, Sauren B, Mohr FW, Walther T, Zickmann B, Iversen S, Felderhoff T, Cartier R, Bonan R. Percutaneous aortic valve replacement for severe aortic stenosis in high-risk patients using the second- and current third-generation self-expanding CoreValve prosthesis: device success and 30-day clinical outcome. J Am Coll Cardiol. 2007 Jul 3;50(1):69-76. doi: 10.1016/j.jacc.2007.04.047. Epub 2007 Jun 6. PMID 17601548

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medtronic CoreValve® System Implantation
Started | 634
Completed | 481
Not Completed | 153
Not completed — Death | 113
Not completed — Withdrawal by Subject | 40

BASELINE CHARACTERISTICS:
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.1 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281
  Male | 353
Region of Enrollment [Number; unit: participants]
  New Zealand | 111
  Australia | 523

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) Rate
Description: Defined as a composite of all cause death, myocardial infarction(MI) (Q-wave & non-Q-wave), stroke, and re-intervention (defined as any emergent cardiac surgery or percutaneous re-intervention catheter procedure that repairs, otherwise alters or adjusts or replaces a previously implanted valve)
Time Frame: 30 days
Measure: Number; unit: probability of events at 30 days
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
probability of events at 30 days | 0.099

2. Primary Outcome: Percentage of Participants With Overall Device Success
Description: * Vascular access, delivery and deployment of the device, and retrieval of the delivery system
  * Correct position of the device in the proper anatomical location (placement in the annulus with no impedance on device function)
  * Intended performance of the prosthetic valve (aortic valve area > 1.2 cm2 (by echocardiography using the continuity equation) and mean aortic valve gradient < 20 mmHg, without moderate or severe prosthetic valve aortic regurgitation)
  * Only one valve implanted
  * No occurrence of in-hospital MACCE
Time Frame: 24-48 hours after the procedure or before the discharge
Measure: Number; unit: % of participants with device success
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
% of participants with device success | 52.6

3. Primary Outcome: Cardiac-related Death
Description: Defined as all death resulting from a cardiac cause or complications of a cardiac procedure and / or death of an unknown cause; this category includes valve-related deaths and non-valve-related cardiac deaths (e.g. congestive heart failure, acute myocardial infarction, documented fatal arrhythmias).
Time Frame: 30 days
Measure: Number; unit: probability of events at 30 days
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
probability of events at 30 days | 0.035

4. Secondary Outcome: All-Cause Mortality
Description: is defined per Valve Academic Research Consortium-1 consensus document (VARC-1), including Cardiovascular and non-cardiovascular mortality.
Time Frame: 30 days
Measure: Number; unit: probability of events at 30 days
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
probability of events at 30 days | 0.038

5. Secondary Outcome: Myocardial Infarction
Description: Included Q-wave and non-Q-wave.
Time Frame: 30 days
Measure: Number; unit: probability of events at 30 days
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
probability of events at 30 days | 0.021

6. Secondary Outcome: Stroke
Description: Is a neurological deficit lasting more than 24 hours, or lasting 24 hours or less with a brain imaging study showing infarction.
Time Frame: 30 days
Measure: Number; unit: probability of events at 30 days
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
probability of events at 30 days | 0.043

7. Secondary Outcome: Re-intervention
Description: Any emergent surgical or percutaneous interventional catheter procedure that repairs, otherwise alters or adjusts, or replaces a previously implanted valve.
Time Frame: 30 days
Measure: Number; unit: probability of events at 30 days
Arm/Group | Medtronic CoreValve® System Implantation
Number analyzed (Participants) | 634
probability of events at 30 days | 0.019

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Medtronic CoreValve® System Implantation
Serious Adverse Events (participants affected / at risk) | 534/634
Other Adverse Events (participants affected / at risk) | 583/634
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic CoreValve® System Implantation (N=634)
Atrioventricular block (Cardiac disorders) | 125 (126)
Cardiac failure congestive (Cardiac disorders) | 84 (120)
Anaemia (Blood and lymphatic system disorders) | 57 (71)
Atrial fibrillation (Cardiac disorders) | 45 (53)
Renal failure (Renal and urinary disorders) | 42 (46)
Pneumonia (Infections and infestations) | 41 (50)
Cerebrovascular accident (Nervous system disorders) | 40 (42)
Angina Pectoris (Cardiac disorders) | 31 (37)
Cardiac failure (Cardiac disorders) | 31 (35)
Myocardial infarction (Cardiac disorders) | 31 (35)
Paravalvular aortic regurgitation (Cardiac disorders) | 30 (30)
Hypotension (Vascular disorders) | 27 (30)
Bundle branch block left (Cardiac disorders) | 23 (23)
Haematoma (Vascular disorders) | 22 (22)
Bradycardia (Cardiac disorders) | 19 (19)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 19 (20)
Sepsis (Infections and infestations) | 18 (20)
Urinary tract infection (Infections and infestations) | 17 (17)
Non-cardiac chest pain (General disorders) | 15 (18)
Vascular access site pseudoaneurysm (General disorders) | 15 (16)
Fall (Injury, poisoning and procedural complications) | 14 (15)
Fractured neck of femur (Injury, poisoning and procedural complications) | 14 (14)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 13 (13)
Syncope (Nervous system disorders) | 13 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (15)
Cellulitis (Infections and infestations) | 12 (14)
Gastrointestinal bleed (Gastrointestinal disorders) | 11 (14)
Transient ischaemic attack (Nervous system disorders) | 11 (12)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 (13)
Rectal haemorrhage (Gastrointestinal disorders) | 10 (10)
Multi-organ disorder (General disorders) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (12)
Cardiac tamponade (Cardiac disorders) | 9 (9)
Cardiogenic shock (Cardiac disorders) | 9 (9)
Ventricular failure (Cardiac disorders) | 9 (9)
Infection (Infections and infestations) | 9 (10)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 9 (9)
Haemoglobin decreased (Investigations) | 9 (9)
Paravalvular leak (Product Issues) | 9 (9)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Postural hypotension (Vascular disorders) | 9 (10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 8 (9)
Cardiac arrest (Cardiac disorders) | 8 (8)
Sinus node dysfunction (Cardiac disorders) | 8 (8)
Melaena (Gastrointestinal disorders) | 8 (9)
Diverticulitis (Infections and infestations) | 8 (8)
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 8 (8)
Femoral artery dissection (Vascular disorders) | 8 (8)
Ventricular tachycardia (Cardiac disorders) | 7 (7)
Confusional state (Psychiatric disorders) | 7 (7)
Haematuria (Renal and urinary disorders) | 7 (7)
Left ventricular failure (Cardiac disorders) | 6 (6)
Fatigue (General disorders) | 6 (6)
Hospital acquired pneumonia (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 6 (7)
Pelvic fracture (Injury, poisoning and procedural complications) | 6 (6)
Iliac artery perforation (Vascular disorders) | 6 (6)
Asystole (Cardiac disorders) | 5 (5)
Atrial flutter (Cardiac disorders) | 5 (6)
Gastrointestinal polyp (Gastrointestinal disorders) | 5 (6)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 5 (6)
Lower respiratory tract infection (Infections and infestations) | 5 (6)
Vascular access site infection (Infections and infestations) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Gout (Metabolism and nutrition disorders) | 5 (6)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (7)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6)
Urinary retention (Renal and urinary disorders) | 5 (5)
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 5 (9)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Hypertension (Vascular disorders) | 5 (5)
Cardiac failure chronic (Cardiac disorders) | 4 (4)
Coronary artery disease (Cardiac disorders) | 4 (4)
Ischaemic mitral regurgitation (Cardiac disorders) | 4 (5)
Pericardial effusion (Cardiac disorders) | 4 (5)
Ventricular fibrillation (Cardiac disorders) | 4 (4)
Right inguinal hernia (Gastrointestinal disorders) | 4 (4)
Upper gastrointestinal bleeding (Gastrointestinal disorders) | 4 (4)
Pain (General disorders) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 4 (4)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 4 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (5)
Dizziness (Nervous system disorders) | 4 (5)
Presyncope (Nervous system disorders) | 4 (4)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hip arthroplasty (Surgical and medical procedures) | 4 (4)
Arterial stenosis (Vascular disorders) | 4 (5)
Haemorrhage (Vascular disorders) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 3 (3)
Cardiac perforation (Cardiac disorders) | 3 (3)
Intracardiac thrombus (Cardiac disorders) | 3 (3)
Pulseless electrical activity (Cardiac disorders) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 3 (3)
Ventricular arrhythmia (Cardiac disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (3)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 3 (3)
Gastric ulcer (Gastrointestinal disorders) | 3 (3)
Gastrointestinal ischaemia (Gastrointestinal disorders) | 3 (3)
Chest pain (General disorders) | 3 (3)
Dysplasia (General disorders) | 3 (3)
Oedema (General disorders) | 3 (4)
Adverse drug reaction (Immune system disorders) | 3 (3)
Bronchitis (Infections and infestations) | 3 (3)
Community acquired pneumonia (Infections and infestations) | 3 (3)
Endocarditis (Infections and infestations) | 3 (3)
Endocarditis viral (Infections and infestations) | 3 (3)
Febrile infection (Infections and infestations) | 3 (3)
Gastroenteritis (Infections and infestations) | 3 (4)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 3 (3)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 3 (3)
Vascular access site complication (Injury, poisoning and procedural complications) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Lethargy (Nervous system disorders) | 3 (3)
Delirium (Psychiatric disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Embolism arterial (Vascular disorders) | 3 (3)
Vascular dissection (Vascular disorders) | 3 (3)
Bifascicular block (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (3)
Systolic dysfunction (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Bilateral inguinal hernia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 2 (2)
Rectal polyp (Gastrointestinal disorders) | 2 (2)
Ulcer (General disorders) | 2 (2)
Unknown cause of death (General disorders) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 2 (2)
Infective exacerbation of bronchiectasis (Infections and infestations) | 2 (2)
Viral infection (Infections and infestations) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2)
Traumatic haemothorax (Injury, poisoning and procedural complications) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 2 (2)
Carotid artery stenosis (Nervous system disorders) | 2 (2)
Neuritis (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Artery dissection (Vascular disorders) | 2 (2)
Femoral artery perforation (Vascular disorders) | 2 (2)
Ischaemia (Vascular disorders) | 2 (2)
Vascular occlusion (Vascular disorders) | 2 (2)
Intracardiac thrombus (Vascular disorders) | 2 (2)
Anaemia of chronic disease (Blood and lymphatic system disorders) | 1 (1)
Anaemia postoperative (Blood and lymphatic system disorders) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1)
Atrioventricular dissociation (Cardiac disorders) | 1 (1)
Aystole (Cardiac disorders) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Diastolic dysfunction (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Left ventricular enlargement (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Trifascicular block (Cardiac disorders) | 1 (1)
Ventricular septal defect acquired (Cardiac disorders) | 1 (1)
Product issues (Product Issues) | 1 (1)
Adrenal mass (Endocrine disorders) | 1 (1)
Diabetes mellitus inadequate control (Endocrine disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Swollen tear duct (Eye disorders) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Volvulus of small bowel (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Complication of device insertion (General disorders) | 1 (1)
Crepitations (General disorders) | 1 (1)
Device embolisation (General disorders) | 1 (2)
Fever of unknown origin (General disorders) | 1 (1)
General system disorders (General disorders) | 1 (1)
Ischaemic ulcer (General disorders) | 1 (1)
Necrosis (General disorders) | 1 (1)
Perforation (General disorders) | 1 (1)
Puncture site haemorrhage (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Bacterial sepsis (Infections and infestations) | 1 (1)
Brain abscess (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Endophthalmitis (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Septic arthritis streptococcal (Infections and infestations) | 1 (1)
Sinusitis fungal (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertibral fracture L2 (Injury, poisoning and procedural complications) | 1 (1)
Oesophageal mucosal tear (Injury, poisoning and procedural complications) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Periprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory distress (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Transurethral resection syndrome (Injury, poisoning and procedural complications) | 1 (1)
Vascular access site dissection (Injury, poisoning and procedural complications) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Colonoscopy (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
False positive investigation result (Investigations) | 1 (1)
International normalised ratio increased (Investigations) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
White blood cell analysis abnormal (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endocrine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Brain injury (Nervous system disorders) | 1 (1)
Brain stem embolism (Nervous system disorders) | 1 (1)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1)
Cluster headache (Nervous system disorders) | 1 (1)
Dementia (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hemiplegia (Nervous system disorders) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Pneumonia (Nervous system disorders) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)
Device pacing issue (Product Issues) | 1 (1)
Delusion (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Psychogenic seizure (Psychiatric disorders) | 1 (2)
Social avoidant behaviour (Psychiatric disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder stenosis (Renal and urinary disorders) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Hypotonic urinary bladder (Renal and urinary disorders) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1)
Renal ischaemia (Renal and urinary disorders) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1)
Uraemia odour (Renal and urinary disorders) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiolitis obliterans with organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pyroderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1)
Bladder neck operation (Surgical and medical procedures) | 1 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 1 (1)
Cardiac rehabilitation therapy (Surgical and medical procedures) | 1 (1)
Hospitalisation (Surgical and medical procedures) | 1 (1)
Joint surgery (Surgical and medical procedures) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Left atrial appendage occlusion (Surgical and medical procedures) | 1 (1)
Pacemaker generated rhythm (Surgical and medical procedures) | 1 (1)
Peripheral endarterectomy (Surgical and medical procedures) | 1 (1)
Rectal prolapse repair (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Aortic dissection (Vascular disorders) | 1 (1)
Aortic rupture (Vascular disorders) | 1 (1)
Arterial haemorrhage (Vascular disorders) | 1 (1)
Basal ganglia haemorrhage (Vascular disorders) | 1 (1)
Femoral artery stenosis (Vascular disorders) | 1 (1)
Iliac artery rupture (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Raynaud's phenomenon (Vascular disorders) | 1 (1)
Subclavian artery perforation (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm ruptured (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medtronic CoreValve® System Implantation (N=634)
Bundle branch block left (Cardiac disorders) | 326 (334)
Vascular access site haematoma (Injury, poisoning and procedural complications) | 92 (104)
Atrioventricular block (Cardiac disorders) | 81 (87)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 63 (69)
Atrial fibrillation (Cardiac disorders) | 55 (57)
Haemoglobin decreased (Investigations) | 49 (51)
Pyrexia (General disorders) | 45 (45)
Hypotension (Vascular disorders) | 44 (44)
Anaemia (Blood and lymphatic system disorders) | 41 (43)
Urinary tract infection (Infections and infestations) | 40 (41)
Haematoma (Vascular disorders) | 39 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes